CLINICAL TRIAL: NCT02104180
Title: Evaluation of the Non-inferiority of TulleGras M.S.® Versus Urgotul® in Pain Associated With Removal of Wound Dressing During Care of Venous Leg Ulcer. An Open-label, Multicenter, Randomized, Controlled, Crossover Study With Blinded Reading of Healing Criteria.
Brief Title: Evaluation of Pain Associated With the Removal of Wound Dressing During Care of Venous Leg Ulcer. Comparison of the Efficacy and Safety of Two Dressings Urgotul and TulleGras
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mylan Inc. (Industry)
Collaborators: CEN Biotech (Industry)
Responsible Party: Sponsor
Organization: Viatris Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: LINE4001; 2013-A01285-40 (Other: ANSM (French Health Agency) Registry number for biomedical research)
Record Dates: First submitted 2014-02-27; First posted 2014-04-04 (Estimated); Results first posted 2019-06-10 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2017-03

CONDITIONS: Venous Leg Ulcer
Keywords: non-inferiority; randomized; TulleGras; Urgotul; pain; venous leg ulcer; healing
MeSH Terms: conditions — Varicose Ulcer; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TulleGras M.S. (Active Comparator)
  Interventions: Device: TulleGras M.S.
- Urgotul (Active Comparator)
  Interventions: Device: Urgotul

INTERVENTIONS:
Device: Urgotul — sterile, hydrocolloid dressing, that consist of a polyester fabric coated with hydrocolloid particles and vaseline
  Arms: Urgotul
Device: TulleGras M.S. — Sterile dressing that consists of viscose tissue coated with mineral vaseline
  Arms: TulleGras M.S.

SUMMARY:
Evaluation of the non-inferiority of TulleGras M.S.® versus Urgotul® in pain associated with removal of wound dressing during care of venous leg ulcer

ELIGIBILITY:
Inclusion Criteria:

* Subject informed of the objectives, purpose, details and constraints of the study and who has given his/her written informed consent.
* Male or female subject.
* Subject at least 45 years of age.
* Subject presenting with an open venous leg ulcer.
* Age of venous leg ulcer between 1 month and 12 months inclusive at the Inclusion Visit (Visit 1).
* Venous leg ulcer whose area is between 4 cm2 and 50 cm2 inclusive at the Inclusion Visit (Visit 1).
* Venous leg ulcer in the granulation phase over 50% of its area at the Inclusion Visit (Visit 1);

Exclusion Criteria:

Related to the disease studied:

* Venous leg ulcer for which surgery is indicated or for which a surgical procedure is planned within twelve weeks of inclusion in the study (Visit 1).
* Venous leg ulcer at start of cleaning phase;
* Fibrinous and dry ulcer (non exudative wound) or on the contrary highly exudative and/or hemorrhagic.
* Venous leg ulcer with signs of critical colonization or clinically infected.
* Cancerous venous leg ulcer.

Related to the subject:

* Subject presenting with a serious systemic disease, which may lead to premature termination of the study before the end of the twelve weeks of treatment of the Follow up Period.
* Subject with a medical history or a significant disease revealed by history which can limit his/her participation or prevent the subject from completing the study.
* Subject presenting with a progressive neoplasm, treated with radiotherapy or chemotherapy or immunosuppressant therapy or high-dose corticosteroids.
* Subject who underwent surgery directly related to his/her venous disease during the two months prior to Inclusion Visit (Visit 1).
* Subject with poorly controlled diabetes.
* Subject who presented with a deep venous thrombosis during the 3 months prior to Inclusion Visit (Visit 1).
* Subject confined to bed.
* Woman of child-bearing potential (NOT postmenopausal for at least 24 months or NOT surgically sterilized (tubal ligation) or NOT hysterectomized) who is NOT routinely using adequate and efficient hormonal contraception or barrier method (intrauterine device, diaphragm, combination of condom and spermicide) prior to and during the trial.
* Subject whose ankle has a circumference, measured at the Inclusion Visit (Visit 1), greater than 32 cm (> 32 cm).
* Subject presenting with symptomatic or asymptomatic peripheral arterial disease, particularly with a distal systolic pressure index, measured at the Inclusion Visit (Visit 1), ≤0.8 or ≥1.3.
* Subject with a history of allergic reaction(s) to one of the different components of the dressings or with a contra-indication to the use of one of these dressings.
* Known history of alcohol abuse or drug abuse.
* Subject linguistically or psychologically unable to understand the information given and to provide informed consent.
* Subject participating in or who participated in another clinical study within 4 weeks prior to the Inclusion Visit (Visit 1).
* Subject not covered by or not a beneficiary of the Social Security system.
* Subject deprived of his freedom as the result of a legal or administrative decision or subject to legal guardianship.
* Any other reason, in the investigator's opinion, that prohibits the inclusion of the subject into the study.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2014-02; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roger Lesaunier, MD, Study Director — Mylan Inc.
Locations (27):
- France (27):
  - Research Facility ID ORG-001183, Angoulème
  - Research Facility ID ORG-000857, Annecy
  - Research facility ID ORG-000853, Asnières
  - Research facility ID ORG-000981, Beaune
  - Research Facility ID ORG-000844, Boulogne-sur-Mer
  - Research Facility ID ORG-000869, Bourgoin
  - Research facility ID ORG-001215, Brest
  - Research Facility ID ORG-001181, Figeac
  - Research facility ID ORG-001081, Grenoble
  - Research Facility ID ORG-000850, Hazebrouck
  - Research facility ID ORG-000855, Lattes
  - Research Facility ID ORG-000859, Laxou
  - Research Facility ID ORG-000830, Lyon
  - Research facility ORG-001362, Melun
  - Research Facility ID ORG-001182, Montpellier
  - Research facility ID ORG-000836, Nancy
  - Research facility ORG-001361, Nantes
  - Research facility ID ORG-000831, Paris
  - Research Facility ID ORG-000832, Paris
  - Research facility ID ORG-000856, Pézenas
  - Research facility ID ORG-001082, Saint-Aubin-sur-Scie
  - Research facility ID ORG-000865, Saint-Maur
  - Research facility ID ORG-000845, Tarare
  - Research facility ID ORG-001216, Toulon
  - Research facility ID ORG-001083, Toulouse
  - Research Facility ID ORG-000862, Tours
  - Research facility ID ORG-000835, Vincennes

RESULTS

PARTICIPANT FLOW:
Groups:
- TulleGras MS - Urgotul: Cross-over period: one dressing of TulleGras M.S. for two days, then one dressing of Urgotul for two days; Follow-up period: Urgotul for a maximum duration of 12 weeks
- Urgotul - TulleGras MS: Cross-over period: one dressing of Urgotul for two days, then one dressing of TulleGras M.S. for two days; Follow-up period: TulleGras M.S. for a maximum duration of 12 weeks
Period: Overall Study
Arm/Group | TulleGras MS - Urgotul | Urgotul - TulleGras MS
Started | 31 | 31
Completed | 30 | 31
Not Completed | 1 | 0
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Urgotul - TulleGras M.S.: Cross-over period: one dressing of Urgotul for two days, then one dressing of TulleGras M.S. for two days; Follow-up period: TulleGras M.S. for a maximum duration of 12 weeks
- Total: Total of all reporting groups
Arm/Group | TulleGras MS - Urgotul | Urgotul - TulleGras M.S. | Total
Number analyzed (Participants) | 31 | 31 | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 78.3 (10.5) | 77.5 (13.7) | 77.9 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 20 | 44
  Male | 7 | 11 | 18
Region of Enrollment [Count of Participants; unit: Participants]
  France | 31 | 31 | 62

OUTCOME MEASURES:

1. Primary Outcome: Pain Intensity at Removal of the Primary Dressing, Evaluated by the Subject Just After Removal
Description: Pain intensity experienced by subjects associated to removal of each study primary dressings during the care, assessed at of the Cross-over Period on a visual analogue scale (VAS). The VAS was provided as a 100 mm, non-graduated horizontal line, with extremities indicating " no pain " (0) and " extreme pain " (100). The subject responded by drawing a vertical line to assess the pain intensity he/she experienced at the time of removal of the primary wound dressing.
Time Frame: at the time of dressing removal on Day 2 (Visit 2) and Day 4 (Visit 3)
Population: Per protocol
Measure: Mean (Standard Deviation); unit: units on a scale: 0-100 mm
Arm/Group | TulleGras M.S. | Urgotul
Number analyzed (Participants) | 61 | 61
units on a scale: 0-100 mm | 11.9 (15.6) | 11.7 (16.7)
Statistical Analysis 1: Comparison: TulleGras M.S. vs Urgotul; Test type: Non-Inferiority — An estimate of the difference between the pain felt by patient during the two dressings removals along with a 95% confidence interval (CI) has been derived. If the upper limit of the confidence interval was less than 13 mm, clinical non-inferiority of Tulle Gras versus Urgotul has been demonstrated; Mean Difference (Final Values) = 0.26, 95% CI 2-sided [-1.339 to 1.864] — The pain intensity has been analyzed using analysis of variance (ANOVA). The model for this cross-over study included sequence, period and treatment as fixed effects and subject within sequence as random effect

ADVERSE EVENTS:
Time Frame: AE collection during the whole study + 30 days following last Patient visit
Arm/Group | TulleGras MS - Urgotul | Urgotul - TulleGras MS
All-Cause Mortality (participants affected / at risk) | 0/31 | 2/31
Serious Adverse Events (participants affected / at risk) | 3/31 | 7/31
Other Adverse Events (participants affected / at risk) | 4/31 | 3/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TulleGras MS - Urgotul (N=31) | Urgotul - TulleGras MS (N=31)
FLARE OF POLYARTHRITIS RHEUMATICA ACUTA (Musculoskeletal and connective tissue disorders) | 0 | 1
VENOUS ULCERATION (Skin and subcutaneous tissue disorders) | 1 | 1
INTERNATIONAL NORMALIZED RATIO ABNORMAL (Investigations) | 0 | 1
BASOCELLULAR CARCINOMA (Skin and subcutaneous tissue disorders) | 0 | 1
OSTEITIS (Musculoskeletal and connective tissue disorders) | 0 | 1
PERIPHERAL VASCULAR DISEASE (Vascular disorders) | 1 | 0
AGGRAVATION OF SKIN ULCER (Skin and subcutaneous tissue disorders) | 1 | 0
ACUTE RESPIRATORY DISTRESS SYNDROME (Respiratory, thoracic and mediastinal disorders) | 0 | 1 — Death after D60 during the study.
DEATH BY CANCER AGGRAVATION (General disorders) | 0 | 1 — D30 after the end of study (LPLV)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TulleGras MS - Urgotul (N=31) | Urgotul - TulleGras MS (N=31)
VENOUS ULCERATION (Skin and subcutaneous tissue disorders) | 0 | 2
ECZEMA (Skin and subcutaneous tissue disorders) | 0 | 1
LEG PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0
TORTICOLLIS (Musculoskeletal and connective tissue disorders) | 1 | 0
CONTACT DERMATITIS (Skin and subcutaneous tissue disorders) | 1 | 0
POPLITEAL CYST (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No